CLINICAL TRIAL: NCT02318173
Title: International Observational E-Registry on the Use of Dilapan-S / Dilasoft Osmotic Dilators for Cervical Ripening Prior to Labour Induction
Brief Title: Dilapan-S/Dilasoft E-Registry in Induction of Labor
Acronym: DSREGISTRYIL
Status: Completed | Type: Observational
Sponsor: Medicem International CR s.r.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: DIS-2014-009
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Labour Onset and Length Abnormalities; Labor; Forced or Induced, Affecting Fetus or Newborn
Keywords: Cervical dilatation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Dilapan-S — Synthetic osmotic dilators Dilapan-S, Dilasoft for cervical ripening prior to induction of labor in women with unfavourable cervix
  Other Names: Dilasoft

SUMMARY:
International Observational E-Registry on the use of DILAPAN-S® osmotic dilator / DILASOFT® osmotic dilator for cervical ripening prior to labour induction.

DETAILED DESCRIPTION:
International Observational E-Registry to monitor current common clinical practice of use of Dilapan-S / Dilasoft for cervical ripening and following procedures of labour induction with the main focus on the duration of induced labor procedure .

ELIGIBILITY:
Inclusion Criteria:

* Indication for induction of labor
* Unfavourable cervix

Exclusion Criteria:

* Presence of overt genital tract infection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients in whom the use of osmotic dilators Dilapan-S or Dilasoft is indicated by the Investigator after a thorough Medical examination will be included in the study unless that the patient disagree.
Sampling Method: Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Duration of Dilapan-S/Dilasoft insertion | max. up to 24 hrs; estimated average 12 hrs)
  duration of cervical ripening
Induction - delivery interval | estimated maximum up to 72 hrs
  Overall duration of induced labor procedure
Rate of vaginal deliveries within 24 hours | up to 24 hrs
  Rate of vaginal deliveries achieved within 24 hours from the beginning of induced labor procedure

SECONDARY OUTCOMES:
Type of osmotic dilator used: Dilapan-S or Dilasoft | up to 24 hrs; estimated average 12 hrs
Number of dilators inserted | up to 24 hrs; estimated average 12 hrs
Bishop Score increase after extraction of osmotic dilators | up to 24 hrs; estimated average 12 hrs
Complications during pre-induction | up to 24 hrs; estimated average 12 hrs
  uterine contractions, uterine hypersensitivity, effect on the foetus
Agents / procedures used for induction of labour, if any | estimated maximum up to 72 hrs
  which, total dosage
% of spontaneous vaginal deliveries following immediately after pre-induction | up to 24 hrs
% of total spontaneous vaginal deliveries | estimated maximum up to 72 hrs
% of instrumented vaginal deliveries | estimated maximum up to 72 hrs
% of Caesarean sections | estimated maximum up to 72 hrs
Foetal status | 0, 5 and 10 minutes after delivery (estimated maximum up to 72 hrs)
  Apgar score at 0, 5 and 10 minutes after delivery, venous and arterial cord pH and base excess measurements
Maternal infectious complication and its relation to the use of Dilapan-S/Dilasoft | up to 72 hrs; Complications, if any, will be followed-up until stable situation has been reached.
  Clinical signs of maternal infection found at patient´s examination are defined as follows:
  1. Body temperature > 37.8°C
  2. Increased pain
  3. Other overt clinical signs of infection e.g. vaginal discharge
     Laboratory test results that need to be correlated with clinical signs of infection:
  4. CRP levels > 8 mg/l
  5. Leukocyte count > 18 x 109/l
  6. Positive microbiological testing
Neonatal infectious complication and its relation to the use of Dilapan-S/Dilasoft | up to 72 hrs; Complications, if any, will be followed-up until stable situation has been reached.
  Clinical signs of neonatal infection found at patient´s examination are defined as follows:
  1. Body temperature > 37.8°C
  2. Increased pain
  3. Other overt clinical signs of infection e.g. vaginal discharge
     Laboratory test results that need to be correlated with clinical signs of infection:
  4. CRP levels > 8 mg/l
  5. Leukocyte count > 18 x 109/l
  6. Positive microbiological testing

CONTACTS AND LOCATIONS:
Overall Officials: Lars Hellmeyer, Doz, MD, Principal Investigator — Vivantes Klinikum im Friedrichshain, Berlin, Germany; Franz Bahlman, Doz, MD, Principal Investigator — Buerger Hospital, Frankfurt am Main, Germany; Janesh Gupta, MD, FRCOG, Study Chair — Birmingham Women´s Hospital, Birmingham, UK; Petr Janku, MD, Principal Investigator — Masaryk University Hospital, Brno, Czech Republic; Jozef Zahumensky, Doc, MD, Principal Investigator — University Hospital, Trnava, Slovakia; Oleg Baev, MD, PhD, Principal Investigator — Federal State Budget Institution "Research Center for Obstetrics, Gynecology and Perinatology" of the Ministry of Healthcare of Russian Federation, Moscow, RUS; Antonio Saad, MD, PhD, Principal Investigator — University of Texas Medical Branch Galveston, TX, US; Amitasrigowri Murthy, MD, PhD, Principal Investigator — Bellevue Hospital, New York City, NY, US; Amita Suneja, Prof, MD, Principal Investigator — Guru Teg Bahadur Hospital, New Delhi, India; Usha Vishwanath, MD, Principal Investigator — Sri Ramachandra Medical Center, Chennai, India; Anisha Gala, MD, Principal Investigator — Fernandez Hospital, Hyderabad, India
Locations (11):
- United States (2):
  - Bellevue Hospital, New York, New York
  - University of Texas Medical Branch Galveston, Galveston, Texas
- Masaryk University, Brno, Czechia
- Germany (2):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Buerger Hospital, Frankfurt am Main
- India (3):
  - Guru Teg Bahadur Hospital, New Delhi, National Capital Territory of Delhi
  - Sri Ramachandra Medical Center, Chennai, Tamil Nadu
  - Fernandez Hospital, Hyderabad, Telangana
- Federal State Budget Institution "Research Center for Obstetrics, Gynecology and Perinatology" of the Ministry of Healthcare of Russian Federation, Moscow, Russia
- University Hospital Trnava, Trnava, Slovakia
- Birmingham Women´s Hospital, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Sanchez-Ramos L. Induction of labor. Obstet Gynecol Clin North Am. 2005 Jun;32(2):181-200, viii. doi: 10.1016/j.ogc.2004.12.004. PMID 15899354
- [Background] Tenore JL. Methods for cervical ripening and induction of labor. Am Fam Physician. 2003 May 15;67(10):2123-8. PMID 12776961
- [Background] Ten Eikelder ML, Neervoort F, Oude Rengerink K, van Baaren GJ, Jozwiak M, de Leeuw JW, de Graaf I, van Pampus MG, Franssen M, Oudijk M, van der Salm P, Woiski M, Pernet PJ, Feitsma AH, van Vliet H, Porath M, Roumen F, van Beek E, Versendaal H, Heres M, Mol BW, Bloemenkamp KW. Induction of labour with a Foley catheter or oral misoprostol at term: the PROBAAT-II study, a multicentre randomised controlled trial. BMC Pregnancy Childbirth. 2013 Mar 19;13:67. doi: 10.1186/1471-2393-13-67. PMID 23506128
- [Background] Jozwiak M, ten Eikelder M, Oude Rengerink K, de Groot C, Feitsma H, Spaanderman M, van Pampus M, de Leeuw JW, Mol BW, Bloemenkamp K; PROBAAT Study Group. Foley catheter versus vaginal misoprostol: randomized controlled trial (PROBAAT-M study) and systematic review and meta-analysis of literature. Am J Perinatol. 2014 Feb;31(2):145-56. doi: 10.1055/s-0033-1341573. Epub 2013 Apr 5. PMID 23564065
- [Background] Sciscione AC, McCullough H, Manley JS, Shlossman PA, Pollock M, Colmorgen GH. A prospective, randomized comparison of Foley catheter insertion versus intracervical prostaglandin E2 gel for preinduction cervical ripening. Am J Obstet Gynecol. 1999 Jan;180(1 Pt 1):55-60. doi: 10.1016/s0002-9378(99)70149-3. PMID 9914578
- [Background] Cromi A, Ghezzi F, Uccella S, Agosti M, Serati M, Marchitelli G, Bolis P. A randomized trial of preinduction cervical ripening: dinoprostone vaginal insert versus double-balloon catheter. Am J Obstet Gynecol. 2012 Aug;207(2):125.e1-7. doi: 10.1016/j.ajog.2012.05.020. Epub 2012 Jun 1. PMID 22704766
- [Background] Suffecool K, Rosenn BM, Kam S, Mushi J, Foroutan J, Herrera K. Labor induction in nulliparous women with an unfavorable cervix: double balloon catheter versus dinoprostone. J Perinat Med. 2014 Mar;42(2):213-8. doi: 10.1515/jpm-2013-0152. PMID 24096438
- [Background] Lichtenberg ES. Complications of osmotic dilators. Obstet Gynecol Surv. 2004 Jul;59(7):528-36. doi: 10.1097/00006254-200407000-00022. PMID 15199271
- [Background] Chua S, Arulkumaran S, Vanaja K, Ratnam SS. Preinduction cervical ripening: prostaglandin E2 gel vs hygroscopic mechanical dilator. J Obstet Gynaecol Res. 1997 Apr;23(2):171-7. doi: 10.1111/j.1447-0756.1997.tb00828.x. PMID 9158305
- [Derived] Gupta J, Chodankar R, Baev O, Bahlmann F, Brega E, Gala A, Hellmeyer L, Hruban L, Maier J, Mehta P, Murthy A, Ritter M, Saad A, Shmakov R, Suneja A, Zahumensky J, Gdovinova D. Synthetic osmotic dilators in the induction of labour-An international multicentre observational study. Eur J Obstet Gynecol Reprod Biol. 2018 Oct;229:70-75. doi: 10.1016/j.ejogrb.2018.08.004. Epub 2018 Aug 3. PMID 30107363